CLINICAL TRIAL: NCT03892031
Title: Preliminary Study on the Changes of Perioperative Circulatory Function in Patients Undergoing Laparoscopic Radical Cystectomy for Bladder Cancer
Brief Title: Circulatory Function in Laparoscopic Radical Cystectomy for Bladder Cancer
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, DAN HUANG, Principal Investigator, clinical attending in anesthesia department, RenJi Hospital
Other Study IDs: Circulatory function in LRC
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Circulatory Function; Laparoscopic Radical Cystectomy for Bladder Cancer
Keywords: brain natriuretic peptide; pneumoperitoneum; Trendelenburg; circulatory function; laparoscopic radical cystectomy for bladder cancer; central venous pressure; stroke volume variation; transthoracic echocardiography
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To optimize the perioperative management of patients undergoing laparoscopic radical cystectomy(LPC) for bladder cancer through observation of perioperative changes of Brain Natriuretic Peptide(BNP), stroke volume variation(SVV), central venous pressure(CVP) and the use of transthoracic echocardiography(TTE).

DETAILED DESCRIPTION:
Long term pneumoperitoneum and steep trendelenburg in LPC for bladder cancer influence perioperative circulatory function, resulting in a series of pathophysiological changes. BNP is of high sensitivity and specificity in the evaluation of cardiac function. SVV and CVP are dynamic and static indices to predict fluid responsiveness. TTE is a good indicator of volume and cardiac function.Thus, we conducted the trial to assess the perioperative circulatory function in patients undergoing LPC. We hypothesized that long term pneumoperitoneum and steep trendelenburg in LPC for bladder cancer would increase perioperative blood volume and influence cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* undergoing laparoscopic radical cystectomy for bladder cancer
* ASA I-II

Exclusion Criteria:

* Cardiac insufficiency
* Hepatic insufficiency
* Renal insufficiency

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo laparoscopic radical cystectomy for bladder cancer in Renji Hospital
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Brain Natriuretic Peptide(BNP) | before induction (T1), at the end of operation(T2), at 12 hours (T3) and 24 hours (T4) postoperatively
  To observe the change of BNP perioperatively.
Central Venous Pressure(CVP) | before induction (T1),at the end of operation (T2), at 12 hours (T3) and 24 hours (T4) postoperatively
  To observe the change of CVP perioperatively.
Stroke Volume Variation(SVV) | before induction (T1), at the end of operation (T2)
  To observe the change of SVV perioperatively.
Transthoracic Echocardiography | before induction (T1),at the end of operation (T2), at 12 hours (T3) and 24 hours (T4) postoperatively
  To observe the change of End-diastolic volume(EDV) perioperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jie Chen, MS, Study Chair — Renji Hospital, School of Medicine, Shanghai Jiaotong University, China
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, China, Shanghai, Shanghai Municipality, China